CLINICAL TRIAL: NCT00487591
Title: An Evaluation of Simvastatin 20 mg Plus Omacor 4 g Compared to Simvastatin 20 mg Plus Placebo in Subjects With Mixed Dyslipidemia
Brief Title: An Evaluation of Simvastatin Plus Omacor Compared to Simvastatin Plus Placebo in Subjects With Mixed Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Provident Clinical Research (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Kevin C. Maki, PhD, Chief Science Officer, Provident Clinical Research
Other Study IDs: PRV-06009
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Mixed Dyslipidemia
Keywords: cholesterol; dyslipidemia; omega 3
MeSH Terms: conditions — Dyslipidemias | interventions — Omacor; Simvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Simva+Omacor
  Interventions: Drug: Omacor (omega-3-acid ethyl esters)plus simvastatin
- Simva + Placebo
  Interventions: Drug: simvastatin plus placebo

INTERVENTIONS:
Drug: Omacor (omega-3-acid ethyl esters)plus simvastatin — Omacor(omega-3-acid ethyl esters) - 4/g day (4 one gram capsules) simvastatin - 20 mg/day (1 tablet/20 mg)
  Other Names: Lovaza
  Groups: Simva+Omacor
Drug: simvastatin plus placebo — simvastatin 20mg/day (1 tablet 20 mg)plus 4 capsules matching placebo
  Groups: Simva + Placebo

SUMMARY:
The primary objective of this study is to compare the effect of simvastatin plus Omacor to simvastatin plus placebo for lowering non-high density lipoprotein cholesterol in subjects with mixed dyslipidemia.

DETAILED DESCRIPTION:
This trial will utilize a randomized, double-blind, two-period crossover design. At Visit 4 (Week 0), after a 5-week diet lead-in/baseline period, subjects meeting all entry criteria will be randomized to one of two double-blind treatment sequences, simvastatin/Omacor first or simvastatin/placebo first. Each treatment period consists of 6 weeks. After randomization, subjects will self-administer the study drugs once a day in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-79 inclusive
* Fasting, untreated non-high-density lipoprotein cholesterol (non-HDL-C level above ATP III goals
* Fasting, untreated triglyceride (TG) level in the high to very high range
* Provide written informed consent and authorization for protected health information

Exclusion Criteria:

* Pregnancy
* Use of lipid-altering drugs which cannot be stopped
* History of certain cardiovascular conditions or cardiac surgery within the prior 6 months
* Body mass index above 40 kg per square meter
* Allergy or sensitivity to omega-3 fatty acids or to statin drugs
* Poorly-controlled conditions including diabetes, hypertension, or thyroid disease
* Certain muscle, liver, kidney, lung or gastrointestinal conditions
* Certain medications
* Active cancers treated within prior 2 years (except non-melanoma skin cancer)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in non-high-density lipoprotein cholesterol (non-HDL-C) | Baseline to end of treatment

SECONDARY OUTCOMES:
Changes in other lipid and biomarker levels | Baseline through end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Provident Clinical Research

REFERENCES:
- [Result] Maki KC; McKenney JM; Lubin BC; Reeves MS. Lipid effects of prescription omega-3-acid ethyl esters plus simvastatin in subjects with hypertriglyceridemia. FASEB J 2008;22:147.8
- [Result] Maki KC, McKenney JM, Reeves MS, Lubin BC, Dicklin MR. Effects of adding prescription omega-3 acid ethyl esters to simvastatin (20 mg/day) on lipids and lipoprotein particles in men and women with mixed dyslipidemia. Am J Cardiol. 2008 Aug 15;102(4):429-33. doi: 10.1016/j.amjcard.2008.03.078. Epub 2008 May 22. PMID 18678300
- [Result] Maki KC, Lubin BC, Reeves MS, Dicklin MR, Harris WS. Prescription omega-3 acid ethyl esters plus simvastatin 20 and 80 mg: effects in mixed dyslipidemia. J Clin Lipidol. 2009 Feb;3(1):33-8. doi: 10.1016/j.jacl.2008.12.007. Epub 2008 Dec 27. PMID 21291786